CLINICAL TRIAL: NCT06850688
Title: Impact of Ambulatory Continuous Monitoring Using Remote Monitoring Medicine Within Patient's Care Pathway Following Colorectal Surgery - A Multicenter Randomized Study
Brief Title: Impact of Ambulatory Continuous Monitoring Using Remote Monitoring Medicine Within Patient's Care Pathway Following Colorectal Surgery (CONTACT-GRECCAR 21)
Acronym: CONTACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: EPOCA U&I (Industry); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC22_0452; 2024-A01770-47 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2025-02-07; First posted 2025-02-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Surgery; Readmission
Keywords: colorectal surgery; remote monitoring platform; Hospital length of stay; Rehospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional discharge (No Intervention): The patients will be discharged from the hospital through standard discharge procedures. They will be seen on Day 30 during their routine postoperative consultation and then contacted by phone on Day 90. All patients will be required to complete a patient diary from Day 0 to the telephone contact on Day 90 in order to record their healthcare utilization during this period.
- Remote monitoring plateform (Experimental): Patient monitoring via the remote monitoring platform for 30 days after hospital discharge. They will be seen on Day 30 during their routine postoperative consultation and then contacted by phone on Day 90. All patients will be required to complete a patient diary from Day 0 to the telephone contact on Day 90 in order to record their healthcare utilization during this period.
  The qualitative component includes data collection through semi-structured individual interviews with a sample of patients, as well as data collection through focus groups with a sample of healthcare professionals involved in the system.
  Interventions: Device: Remote monitoring platform

INTERVENTIONS:
Device: Remote monitoring platform — EPOCA Intelligence Information System is a remote monitoring plateform. The medical device is used as a SaaS platform with restricted access for healthcare professionals. Patients and their families interact with the medical device via notifications and secure links, upon request. The medical device integrates the use of other medical devices such as oximeters, blood pressure monitors, glucometers, bracelets, etc., which are connected and whose use is also governed by their user manuals and training.
  Patient is monitoring via the remote monitoring platform for 30 days after hospital discharge
  Arms: Remote monitoring plateform

SUMMARY:
The goal of this Clinical Investigation is to evaluate the effectiveness of implementing the discharge protocol of the remote monitoring platform after colorectal surgery in patients at risk of hospital readmission.

Participants will be randomized into either the "30 days of remote monitoring" group or the "conventional discharge" group. The patient returns to the site for their postoperative visit at 30 days and is contacted by phone 90 days after their surgery.

ELIGIBILITY:
Inclusion Criteria :

* Man or woman over 18 years old at the time of the J0 visit,
* Patient who has undergone colorectal surgery not managed on an outpatient basis at the investigator center,
* At least one of the following two criteria:
* Anticipated early discharge (within 24 hours following laparoscopic surgery without diversion and within 5 days following surgery by laparotomy with stoma) for a surgery not managed on an outpatient basis in routine practice,
* Estimated risk of hospital readmission greater than 10% according to the nomogram of Tevis et al. [15], adapted to the postoperative context in digestive surgery (>120 points according to this score).
* Patient affiliated with a health insurance plan,
* Patient who has signed the study consent form.

Exclusion Criteria:

* Discharge to a rehabilitation center requested by the patient,
* Condition managed on an outpatient basis in routine practice for this type of patient,
* Patient eligible for home hospitalization services,
* Suicidal or hetero-aggressive risk in a patient living alone at home
* Homeless patient,
* Pregnant or breastfeeding women,
* Patient under legal guardianship, curatorship, or protected legal status,
* Patient already enrolled in an interventional postoperative follow-up study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-10-17 (Estimated); Study Completion 2026-10-17 (Estimated)

PRIMARY OUTCOMES:
Hospitalization days | 90 days
  Cumulative duration of hospitalization days up to 90 days after the index surgery

SECONDARY OUTCOMES:
Unplanned hospital readmission | 90 days
  Rate of unplanned hospital readmissions with emergency department visits at 90 days
Difference between the initial hospital discharge date and the hospital readmission date | 90 days
  Difference between the initial hospital discharge date and the hospital readmission date (for readmitted patients)
Unplanned consultations | 90 days
  Rate of unplanned consultations at 90 days
Postoperative morbidity | 90 days
  Number of patients presenting a complication out of the total number of patients
Severe postoperative morbidity | 90 days
  Severe postoperative morbidity at 90 days (Clavien-Dindo classification levels 3 and 4)
Visual Analog Scale at Day 3 for preoperative inclusions | Day 3
  Visual Analog Scale at Day 3 for preoperative inclusions. Visual Analog Scale is self-assessment scale (in cm) ranging from 0 (no pain) to 10 (maximum imaginable pain).
Visual Analog Scale at Day 5 for preoperative inclusions | Day 5
  Visual Analog Scale at Day 5 for preoperative inclusions. Visual Analog Scale is self-assessment scale (in cm) ranging from 0 (no pain) to 10 (maximum imaginable pain).
Rate of postoperative ileus at Day 3 for preoperative inclusions | Day 3
  Rate of postoperative ileus at Day 3 for preoperative inclusions
Rate of postoperative ileus at Day 5 for preoperative inclusions | Day 5
  Rate of postoperative ileus at Day 5 for preoperative inclusions
Return to Professional activities | 90 days
  Date of return to professional activities within 90 days
Quality of life questionnaires "Medical Outcomes Study 36-item Short-Form Health Survey" | 30 days
  Quality of life questionnaires"Medical Outcomes Study 36-item Short-Form Health Survey" (SF-36) at 30 days. It consists of 36 questions. Each question is assessed using a Likert scale with 3, 5, or 6 possible response levels. The 8 dimensions also allow for the calculation of two quality-of-life scores: the Physical Composite Score and the Mental Composite Score. The higher the score, the greater the capacity.
Quality of life questionnaires "Medical Outcomes Study 36-item Short-Form Health Survey" | 90 days
  Quality of life questionnaires "Medical Outcomes Study 36-item Short-Form Health Survey " (SF-36) at 90 days. It consists of 36 questions. Each question is assessed using a Likert scale with 3, 5, or 6 possible response levels. The 8 dimensions also allow for the calculation of two quality-of-life scores: the Physical Composite Score and the Mental Composite Score. The higher the score, the greater the capacity.
Quality of life questionnaires EQ-5D | 30 days
  Quality of life questionnaires EQ-5D at 30 days. The questionnaire 5-level EQ-5D version consists of 5 response items indicating an increasing severity of problems in the relevant dimension and a visual analog scale ranging from 0 to 100, assessing overall health status.
Quality of life questionnaires EQ-5D | 90 days
  Quality of life questionnaires EQ-5D at 90 days. The questionnaire 5-level EQ-5D version consists of 5 response items indicating an increasing severity of problems in the relevant dimension and a visual analog scale ranging from 0 to 100, assessing overall health status.
Total cost of the care pathway over 90 days | 90 days
  Costs will be estimated based on hospital stays (initial and any rehospitalizations), outpatient healthcare consumption (limited to medical consultations), and the remote monitoring platform
Patient satisfaction | 30 days
  Likert scale at 30 days to assess the level of patient satisfaction. This questionnaire consists of 3 items (statements) for which the respondent will express their degree of agreement or disagreement. Each statement will be associated with an integer number from 1 to 5 for the quantitative analysis of the data. The final score on this scale will therefore range between 3 and 15.
Number of days between surgery and the resumption of both gaseous and fecal transit within 90 days | 90 days
  Number of days between surgery and the resumption of both gaseous and fecal transit within 90 days
Number of patients maintained at home but discontinuing the use of the remote monitoring platform system before the end of follow-up | 90 days
  Number of patients maintained at home but discontinuing the use of the remote monitoring platform system before the end of follow-up
The reason for patients remaining at home after discontinuing the use of the remote monitoring platform system before the end of the follow-up | 90 days
  Number of patients maintained at home but discontinuing the use of the remote monitoring platform system before the end of follow-up, along with the reasons
Number of patients managed with the remote monitoring platform system | 90 days
  Number of patients managed with the remote monitoring platform system from the day the discharge criteria were met
Duration of use of remote monitoring plateform | 90 days
  Number of days between returning home with the remote monitoring platform system and the end of follow-up by the remote moinitoring platform
Characteristics of the care provided by the remote monitoring platform system | 90 days
  Characteristics of care provided through the remote monitoring platform system, according to the guidelines
Focus groups | 90 days
  Analysis of data collected through focus groups with professionals involved in the system
Patient and caregiver verbatims | 90 days
  Qualitative aspect : Analysis of patient and caregiver verbatims. Evaluation of the patient's and their caregiver's adherence to the system. The collection and analysis of the experiences of thirty families (one patient + one caregiver) will be conducted using two data collection tools : the diary and the semi-structured interview.
Patient verbatims on the post-operative experience | 90 days
  Qualitative aspect : Analysis of patient verbatims on the post-operative experience. Understanding of the patient's experience, including their feelings and anxiety during the postoperative period. The collection and analysis of the experiences of thirty families (one patient + one caregiver) will be conducted using two data collection tools : the diary and the semi-structured interview.
Healthcare professionals' verbatims | 90 days
  Qualitative aspect : Analysis of healthcare professionals' verbatims. Exploring the social, economic, and geographical inequalities in the use of outpatient and/or early hospital discharge. The experience of healthcare professionals will be collected during four focus groups and will help determine the conditions for the implementation and dissemination of the remote monitoring platform system beyond the partner centers and for other health situations.
Medical-economic endpoint | 90 days
  Medical-economic endpoint : Incremental cost-utility ratio (cost per QALY, Quality-Adjusted Life-Year).

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU Angers, Angers
  - Clinique Tivoli- Ducos, Bordeaux
  - CHU Grenoble, Grenoble
  - Centre Hospitalier Lyon-Sud, Lyon
  - CHU Timone - Assistance publique-Hôpitaux de Marseille, Marseille
  - Hôpital Nord - Assistance publique- Hôpitaux de Marseille, Marseille
  - Institut Paoli Calmettes, Marseille
  - CHU Nantes, Nantes
  - Hôpital de Bicêtre - Assistance Publique Hôpitaux de Paris, Paris
  - Hôpital Saint Antoine - Assistance publique - Hôpitaux de Paris, Paris
  - CHU Rennes, Rennes
  - Clinique Mutualiste de l'estuaire, Saint-Nazaire
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided